CLINICAL TRIAL: NCT01095003
Title: A Phase III Trial of Vinflunine Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer Previously Treated With or Resistant to an Anthracycline and Who Are Taxane Resistant.
Brief Title: Trial of Vinflunine Plus Capecitabine in Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L00070 IN 305 B0; 2008-004171-21 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-29 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — vinflunine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vinflunine plus Capecitabine (Experimental): Patients received (in combination with capecitabine)
  • Vinflunine at the dose of 280 mg/m² and as a 20-minute IV. infusion on day 1 of each cycle repeated every 3 weeks.
  Interventions: Drug: Vinflunine plus Capecitabine
- Capecitabine single-agent (Active Comparator): Capecitabine at the dose of 825mg/m² per os twice per day each morning and each evening for 14 consecutive days beginning on day 1 of each cycle repeated every 3 weeks (self-administered).
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Vinflunine plus Capecitabine — Vinflunine 280mg/m² as a 20-minute i.v. infusion on day 1 of each cycle repeated every 3 weeks
  Capecitabine 825mg/m² per os twice per day for 14 consecutive days starting day 1 of each cycle repeated every 3 weeks
  Other Names: JAVLOR; L00070 IN
  Arms: Vinflunine plus Capecitabine
Drug: Capecitabine — Capecitabine 825mg/m² per os twice per day for 14 consecutive days starting day 1 of each cycle repeated every 3 weeks
  Other Names: XELODA
  Arms: Capecitabine single-agent

SUMMARY:
The increasing use of anthracyclines and taxanes in the adjuvant, neoadjuvant and first-line metastatic settings, led to a raise of patients presenting with metastatic breast cancer after treatment with these agents. Options for the treatment of patients who have progressed after an anthracycline and a taxane are limited. The high level of in-vitro synergy of vinflunine combined with 5-fluorouracil (5-FU) together with the good tolerance and the encouraging response rate observed while combining IV vinflunine to oral capecitabine make it a promising combination to investigate further in a phase III trial. This phase III trial will evaluate the effectiveness and the safety profile of such combination for the treatment of patient with advanced breast cancer previously treated with or resistant to anthracycline and taxane resistant.

DETAILED DESCRIPTION:
This multicentre, open-label, randomised, Phase III study will enrol 764 patients with advanced breast cancer who have previously been treated with or are resistant to an anthracycline and who are taxane resistant. Patients will be randomised in a 1:1 ratio to receive vinflunine plus capecitabine (Arm A) or capecitabine alone (Arm B).

Randomisation will be stratified according to a minimization procedure:

1. Resistance to anthracyclines ("yes" versus "no"), Relapse ≤ 12 months in the adjuvant or neoadjuvant setting or progression ≤ 4 months in the metastatic setting,
2. Karnofsky performance status ("90-100" versus "70-80"),
3. Measurable disease ("yes" versus "no"),
4. The number of prior lines of chemotherapy in the metastatic setting ("0" versus "1" versus "> 1") and,
5. Study site.

Patients randomised in Arm A will receive:

* Vinflunine at the dose of 280 mg/m² on day 1 of each cycle every 3 weeks, over a 20-minute i.v. infusion and,
* Capecitabine which will be self-administered by the patient in an outpatient setting. Patients will take 825 mg/m² twice daily per os for 14 consecutive days beginning on day 1 of each cycle followed by 1 week of rest. A cycle of therapy is defined as 3 weeks.

For patients randomised in Arm B, capecitabine will be self administered by the patient in an outpatient setting. Patients will take 1250 mg/m² twice daily per os for 14 consecutive days beginning on day 1 of each cycle followed by 1 week of rest. A cycle of therapy is defined as 3 weeks.

The doses and timing of treatment will be modified based on toxicities experienced by the patient.

Patients will be assessed for toxicity, tumour response and progression at regular intervals during treatment. Patients will be evaluated for safety if they received any study drug. Laboratory values, adverse events and other symptoms will be graded.

Tumour response, progression-free survival and duration of response will be evaluated for all randomised patients. Tumour assessment is to be performed every 6 weeks (+/- 3 working days) from randomisation (regardless of the timing of treatment cycles) until disease progression is documented. Patients who discontinue protocol treatment for reasons other than disease progression will have tumour assessments every 6 weeks until documented disease progression. Patients may continue to receive additional cycles of therapy until progressive disease or intolerable toxicity.

Quality of Life assessment, will be measured by EORTC QLQ-C30 and QLQ-BR23 questionnaires, which will be completed by patients.

The primary endpoint for the trial is progression free survival calculated from the date of randomization until the date of progression or the date of death whatever the reason of death. The analysis of Progression-Free Survival is planned to take place when 615 progressions or deaths have been observed. One interim safety analysis is planned and will take place when 50 patients of each arm have completed at least one cycle of study treatment. It is anticipated that up to 170 active study centres will participate, and that accrual will be completed in approximately 30 months.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* 21 years of age or older
* histologically/cytologically confirmed carcinoma of the breast
* documented locally recurrent or metastatic disease not amenable to curative surgery or radiotherapy
* either one, two or three prior chemotherapy regimens
* prior treatments including both an anthracycline and a taxane and patient no longer candidate for these drugs
* measurable or non-measurable disease according to RECIST 1.1
* Karnofsky performance score of at least 70 %
* adequate haematological, hepatic and renal functions
* ECG without clinically relevant abnormality

Exclusion Criteria:

* known or clinical evidence of brain metastasis or leptomeningeal involvement
* pulmonary lymphangitis or symptomatic pleural effusion
* any serious, concurrent uncontrolled medical disorder
* history of second primary malignancy
* preexisting motor/sensory peripheral neuropathy
* known history of HIV infection
* prior therapy with capecitabine and/or vinca-alkaloids
* history of severe hypersensitivity to vinca alkaloids and/or to fluoropyrimidine or contra indication to any of these drugs
* known or suspected dihydropyrimidine dehydrogenase (DPD) deficiency
* pregnancy or breast feeding

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude VEDOVATO, Study Director — Pierre Fabre Medicament
Locations (110):
- Argentina (5):
  - Buenos Aires
  - Quilmes
  - Rosario
  - San Martín
  - San Miguel de Tucumán
- Belarus (4):
  - Grodno
  - Homyel
  - Minsk
  - Vitebsk
- Belgium (2):
  - Brussels
  - Liège
- Brazil (4):
  - Curitiba
  - Porto Alegre
  - Santo André
  - São Paulo
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Stara Zagora
- Czechia (2):
  - Brno
  - Jihlava
- Tallinn, Estonia
- France (13):
  - Angers
  - Caen
  - Dijon
  - Le Mans
  - Lorient
  - Lyon
  - Montpellier
  - Nantes
  - Saint-Brieuc
  - Saint-Cloud
  - Saint-Herblain
  - Tours
  - Villejuif
- Hungary (3):
  - Budapest
  - Székesfehérvár
  - Szolnok
- India (10):
  - Aurangabad
  - Bangalore
  - Bhopal
  - Calicut
  - Jaipur
  - Kolkata
  - Mumbai
  - Patna
  - Pune
  - Trivandrum
- Italy (10):
  - Avellino
  - Cagliari
  - Cremona
  - Fabriano
  - Milan
  - Monza
  - Padua
  - Pisa
  - Rozzano
  - Verona
- Mexico (4):
  - Chihuahua City
  - León
  - Mexico City
  - Saltillo
- Poland (6):
  - Bialystok
  - Gdansk
  - Krakow
  - Lodz
  - Lubin
  - Warsaw
- Russia (11):
  - Arkhangelsk
  - Chelyabinsk
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Stavropol
  - Tambov
  - Ufa
  - Vladimir
  - Volgograd
- Serbia (2):
  - Kamenitz
  - Niš
- South Africa (4):
  - Durban
  - Kimberley
  - Pretoria
  - Sandton
- Spain (5):
  - Barcelona
  - Lleida
  - Madrid
  - Oviedo
  - Valencia
- Switzerland (3):
  - Genolier
  - Lausanne
  - Winterthur
- Taiwan (2):
  - Taipei
  - Taoyuan District
- Ukraine (6):
  - Cherkasy
  - Dnipropetrovsk
  - Donetsk
  - Khmelnytskyi
  - Kyiv
  - Simferopol
- United Kingdom (10):
  - Belfast
  - Chelmsford
  - Keighley
  - London
  - Nottingham
  - Peterborough
  - Portsmouth
  - Sheffield
  - Southend-on-Sea
  - Sutton

REFERENCES:
- [Derived] Martin M, Campone M, Bondarenko I, Sakaeva D, Krishnamurthy S, Roman L, Lebedeva L, Vedovato JC, Aapro M. Randomised phase III trial of vinflunine plus capecitabine versus capecitabine alone in patients with advanced breast cancer previously treated with an anthracycline and resistant to taxane. Ann Oncol. 2018 May 1;29(5):1195-1202. doi: 10.1093/annonc/mdy063. PMID 29447329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
Started | 384 | 386
Completed | 0 | 0
Not Completed | 384 | 386

BASELINE CHARACTERISTICS:
Groups:
- Capecitabine Single-agent: Capecitabine 825mg/m² per os twice per day for 14 consecutive days starting day 1 of each cycle repeated every 3 weeks
- Vinflunine Plus Capecitabine: Vinflunine plus Capecitabine: Vinflunine 280mg/m² as a 20-minute i.v. infusion on day 1 of each cycle repeated every 3 weeks
  Capecitabine: Capecitabine 825mg/m² per os twice per day for 14 consecutive days starting day 1 of each cycle repeated every 3 weeks
- Total: Total of all reporting groups
Arm/Group | Capecitabine Single-agent | Vinflunine Plus Capecitabine | Total
Number analyzed (Participants) | 386 | 384 | 770
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 340 | 329 | 669
  >=65 years | 46 | 55 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 386 | 384 | 770
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: PFS is defined as time from date of randomization to date of the first documentation of objective tumor progression (according to the Independent Response Review Committee (IRC) and based on RECIST version 1.1) or death due to any cause.
  The PFS was primarily analysed in the Intent-to-treat (ITT) population. Patients lost to follow-up, or without a known record of progression or death at time of analysis had the progression-free survival censored at the date of last tumour assessment or the date of last contact of a follow-up showing no progression, whichever occurs last.
Time Frame: Baseline up to 2 years 7 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
Number analyzed (Participants) | 384 | 386
Months | 5.6 [5.3 to 6.3] | 4.3 [4.1 to 5.6]
Statistical Analysis 1: Comparison: Vinflunine Plus Capecitabine vs Capecitabine Single-agent; The final analysis of progression free survival was conducted once the required number of events(615 progressions or deaths) was reached.using the IRC assessment of date of progressions following the blinded radiological and clinical review of data. Kaplan-Meier curves and life tables by treatment arm were provided.A stratified Cox proportional model was used to compare the two treatment arms; Test type: Superiority; p = 0.0426, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 0.99]

2. Secondary Outcome: Overall Survival
Description: The overall survival (OS) was defined as the duration between the date of randomisation and the date of death from any cause. The OS analysis was performed in the ITT population and the eligible and per protocol populations once the required number of events (631 deaths) was observed Patients lost to follow-up, or without a known record of death at time of analysis had the OS censored at the date of last contact.
Time Frame: Baseline upto 3 years 10 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
Number analyzed (Participants) | 384 | 386
Months | 13.9 [11.9 to 15] | 11.7 [10.8 to 13.5]
Statistical Analysis 1: Comparison: Vinflunine Plus Capecitabine vs Capecitabine Single-agent; Test type: Superiority; p = 0.7657, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.83 to 1.15]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as documentation of complete or partial response that was subsequently confirmed to first documentation of disease progression or to death due to any cause, whichever occurred first.
Time Frame: Baseline upto 2 years 7 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
Number analyzed (Participants) | 384 | 386
Percent | 22.9 [18.8 to 27.5] | 17.9 [14.2 to 22.1]
Statistical Analysis 1: Comparison: Vinflunine Plus Capecitabine vs Capecitabine Single-agent; Test type: Superiority; p = 0.103, Cochran-Mantel-Haenszel

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate defined (DCR) as the sum of confirmed complete response, confirmed partial response and stabilisation rate.
Time Frame: Baseline up to 2 years 7 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
Number analyzed (Participants) | 384 | 386
Percent | 57.3 [52.2 to 62.3] | 47.9 [42.9 to 53]
Statistical Analysis 1: Comparison: Vinflunine Plus Capecitabine vs Capecitabine Single-agent; Test type: Superiority; p = 0.0089, Cochran-Mantel-Haenszel

5. Secondary Outcome: Duration of Response
Description: Measured from the first time that measurement criteria were first met for objective response (documented CR or PR) until recurrence/progression or death whatever the cause.
Time Frame: Baseline up to 2 years 7 months
Population: ITT
Measure: Median (Full Range); unit: Months
Groups:
- Vinflunine Plus Capecitabine: Patients received (in combination with capecitabine)
  • Vinflunine at the dose of 280 mg/m² and as a 20-minute IV. infusion on day 1 of each cycle repeated every 3 weeks.
  Vinflunine plus Capecitabine: Vinflunine 280mg/m² as a 20-minute i.v. infusion on day 1 of each cycle repeated every 3 weeks
  Capecitabine 825mg/m² per os twice per day for 14 consecutive days starting day 1 of each cycle repeated every 3 weeks
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
Number analyzed (Participants) | 384 | 386
Months | 57.3 [52.2 to 62.3] | 47.9 [42.9 to 53]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported from time of first dose of study treatment up to the end of study period (treatment period + follow-up period) up to 5 years 9 months.
Description: AEs were collected from treated patients who received at least one dose of study treatment (383 patients in each arm). The same event may appear as both an AE and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and as nonserious in another. Specific AE tables were generated separately as per European format.
Arm/Group | Vinflunine Plus Capecitabine | Capecitabine Single-agent
All-Cause Mortality (participants affected / at risk) | 345/384 | 348/386
Serious Adverse Events (participants affected / at risk) | 107/383 | 85/383
Other Adverse Events (participants affected / at risk) | 257/383 | 262/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine Plus Capecitabine (N=383) | Capecitabine Single-agent (N=383)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 9 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Reflux gastric (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 2
Haemoytique anaemia (Blood and lymphatic system disorders) | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Anginal pectoris (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 0
Condition aggravated (General disorders) | 2 | 6
Death (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 1
Injection site extravasation (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi organ failure (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 2
Cholecytitis (Hepatobiliary disorders) | 1 | 0
Cholecystetis acute (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinemai (Hepatobiliary disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiaratory tract infection (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Device occlusion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
ALAT increased (Investigations) | 0 | 1
ASTT increased (Investigations) | 0 | 1
Biopsy (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokaelemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasmprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 | 32
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Coma (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Subarachnoid haemorrrhage (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
PPES (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anal fistula excision (Surgical and medical procedures) | 0 | 1
Bile duct stent insertion (Surgical and medical procedures) | 0 | 1
Central venous catherisation (Surgical and medical procedures) | 2 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1
Surgery (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine Plus Capecitabine (N=383) | Capecitabine Single-agent (N=383)
Neutropenia (Blood and lymphatic system disorders) | 73 | 32
Cardiac disorders (Cardiac disorders) | 28 | 22
Eye disorders (Eye disorders) | 23 | 31
Abdominal pain (Gastrointestinal disorders) | 119 | 78
Abdominal pain upper (Gastrointestinal disorders) | 49 | 21
Constipation (Gastrointestinal disorders) | 108 | 30
Diarrhoea (Gastrointestinal disorders) | 86 | 116
Nausea (Gastrointestinal disorders) | 123 | 97
Stomatitis (Gastrointestinal disorders) | 88 | 41
Vomiting (Gastrointestinal disorders) | 106 | 62
Asthenia (General disorders) | 66 | 39
Fatigue (General disorders) | 111 | 92
Injection site reaction (General disorders) | 63 | 0
Oedema peripheral (General disorders) | 21 | 22
Pyrexia (General disorders) | 46 | 35
Hepatobiliary disorders (Hepatobiliary disorders) | 29 | 20
Infections and infestations (Infections and infestations) | 95 | 90
Weight decreased (Investigations) | 113 | 74
Weight increased (Investigations) | 55 | 48
Anorexia (Metabolism and nutrition disorders) | 63 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 39 | 30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 36 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 23
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 | 33
Dizziness (Nervous system disorders) | 33 | 23
Headache (Nervous system disorders) | 59 | 38
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 19
Insomnia (Psychiatric disorders) | 26 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 | 51
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 3
PPES (Skin and subcutaneous tissue disorders) | 90 | 180
Vascular disorders (Vascular disorders) | 61 | 28

LIMITATIONS AND CAVEATS:
No limitations and caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No